CLINICAL TRIAL: NCT03032146
Title: The Effect of a Cardiac Rehabilitation Program on Active Participation in the Community and Exercise Habits Six Months After a Coronary Event
Brief Title: The Effect of a Cardiac Rehabilitation Program on Active Participation in the Community and Exercise Habits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Menachem Nahir, Cardiologist, MD., HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0180-16-EMC
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Cardiac Event
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: Patients with at least a month of cardiac rehabilitation at The Emek Medical Center, Afula. Rehabilitation includes a multidisciplinary program based on physical exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participation in cardiac rehabilitation (Experimental): Patients with at least a month of cardiac rehabilitation at The Emek Medical Center, Afula. Rehabilitation includes a multidisciplinary program based on physical exercise.
  Interventions: Procedure: Cardiac Rehabilitation
- control (No Intervention): Patients who chose not to participate in the rehabilitation program, despite being offered the option.

INTERVENTIONS:
Procedure: Cardiac Rehabilitation — Cardiac rehabilitation is a multidisciplinary framework which focuses on improving the functioning of heart disease patients to facilitate and optimize the return to a regular routine as early as possible. The rehabilitation program provides the tools for the maintenance of a healthy lifestyle, encouraging participants to take part in recreational activities and includes extending their daily functioning.
  Arms: participation in cardiac rehabilitation

SUMMARY:
The aim of this study is to examine the contribution of a cardiac rehabilitation program on the active participation in daily life six months after an acute coronary event.

100 patients will be recruited for the study, 3-10 months after a myocardial infarction and hospitalization in the Emek Medical Center in Afula, Israel.

50 patients recruited for the study who had participated in cardiac rehabilitation will be the experimental group. 50 patients who have not participated in rehabilitation- will be the control group. The groups will be matched for diagnosis, sex and age. Sociodemographic data on patients will be taken from the medical records of the cardiology department and the Cardiac Rehabilitation Institute of the Emek Medical Center..

Course of study: Participants will sign an informed consent form and fill out questionnaires that evaluate active participation in the community. In addition, the physical function and muscle strength of the participants will be evaluated with designated tests. The duration of each meeting will be 60 minutes.

HYPOTHESES

1. Patients who participate in a cardiac rehabilitation program will exhibit higher indices of participation in the community than patients who do not participate.
2. Patients who participate in a cardiac rehabilitation program will display higher levels of physical activity when compared with patients who do not participate.

DETAILED DESCRIPTION:
Cardiac rehabilitation is a multidisciplinary framework which focuses on improving the functioning of heart disease patients to facilitate and optimize the return to a regular routine as early as possible. The rehabilitation program provides the tools for the maintenance of a healthy lifestyle, encouraging participants to take part in recreational activities and includes extending their daily functioning. (IADL- Instrumental Activities of Daily Living). A sedentary lifestyle is a major risk factor for heart disease. Increased levels of physical activity and an active lifestyle have a beneficial effect on most of the risk factors for the heart and blood vessels, including lipid profile, blood pressure and body composition.

In addition to the purely physical component, active participation in managing the household, returning to work and leisure activities in the community, have a positive impact on the mental state and contribute to the quality of life of cardiac patients.

Few studies address the return to a normal social life, most focus on the return to work. Since most cardiac rehabilitation program participants are pensioners, it is important to examine other aspects of their participation in society and everyday life in order to measure the effectiveness of a cardiac rehabilitation program.

The setting up of an initial interview and approval in principle to take part in the study will be arranged with a telephone call to the potential participant and a date will be determined for the meeting..

The interview will be conducted in the subject's home. The interviewer will make sure that the participant understands and agrees to the terms of the research. The participant then will fill in and sign a consent form giving the hospital authorization to use his personal details and medical data (gender, age, religion, place of residence).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of coronary heart disease in the patient's medical file, age of 18 years or more, hospitalization after an acute coronary event, reading and comprehension in the Hebrew language, fulfillment of all requirements to take part in the cardiac rehabilitation program.

Exclusion Criteria:

* An orthopedic, neurological, psychological or cognitive background that prevents participation in a rehabilitation program or physical activity. Patient's request not to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
ACS- Activity Card Sort | 10 min.
  A questionnaire describing participation in social, instrumental and recreational activities. A questionnaire consisting of 89 sections describing implementation activities sonotosimor activity and participation. 20 clauses describe instrumental activity. 35 clauses describe recreational activity that require minimal physical effort and 17 that require a higher level of effort. 17 additional clauses describe leisure activities.
International Physical Activity Questionnaire-IPAQ | 5 min.
  A self-reporting questionnaire measuring physical activity in 27 sections. The questionnaire examines the duration (in minutes) and frequency (in days) of physical activity during the previous 7 days. Activity is measured in the following areas: work, mobility, home maintenance, sports recreation, and while sitting.

SECONDARY OUTCOMES:
MoCA - Montreal Cognitive Assessment Tool | 10 min.
  Examines various cognitive domains: Attention and concentration, memory, language, and conceptual thinking, calculations, and spatial orientation.
TUG - Timed up and go test | 5 min.
  Evaluates: Mobility, stability, ability to walk and risk of falling in adults. Participants are required to perform a task: "You need to get up from a chair, walk 3 meters quickly and confidently, step over a symbol marked on the floor, turn around, go back and sit down on the chair."
Timed Up and Go dual task - with cognitive task | 5 min.
  A dynamic Test, for the evaluation of performance and the risk of falling, during the dual task. The test simulates the conditions of the natural environment in which a person is required to perform multiple tasks Participants are required to perform a task: "You need to get up from a chair, walk 3 meters quickly and confidently, step over a symbol marked on the floor, turn around, go back and sit down on the chair. While performing the task you need to subtract the number 3 from a random number between 20 and 100".
Grip Strength test | 5 min.
  Testing for an objective and quantitative measure of isometric muscle strength of the hand and forearm muscles. Grip strength that is lower than expected for age has been associated with premature mortality, evolving disability and lengthy rehabilitation after surgery or hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Nahir, Principal Investigator — haemek medical center
Locations (1):
- Ran Vainer, Afula, Israel

IPD SHARING:
Plan to Share IPD: No